CLINICAL TRIAL: NCT05286268
Title: The Role of Ischemia Modified Albumin in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Pagonis Athanasios, Pulmonology resident, Larissa University Hospital
Other Study IDs: 24918
Record Dates: First submitted 2022-03-16; First posted 2022-03-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Ischemia Modified Albumin; IMA; Prognosis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with confirmed COVID-19 disease
  Interventions: Diagnostic Test: Ischemia Modified Albumin
- Control group: Healthy volunteers without any of the exclusion criteria
  Interventions: Diagnostic Test: Ischemia Modified Albumin

INTERVENTIONS:
Diagnostic Test: Ischemia Modified Albumin — Blood sampling at admission for measurement of IMA and suPAR levels and at day 10 from symptom onset (peak of symptoms) for IMA level. Samples will be collected in blood collection tubes containing K2EDTA as anticoagulant and serum separation gel tubes for SuPAR and IMA assays respectively. The samples will be centrifuged (at 3000 x g for 10 minutes) within the first 3 hours of sampling. Then, both plasma and serum samples will be placed in Eppendorf tubes and stored at -80oC. IMA levels will be determined according to the principles of the ACB assay, using the commercially available "Ischemia Modified Albumin Assay Kit" method (Abbexa LTD, Cambridge, UK), on the Architect c8000 automatic analytical system (Abbott, USA). SuPAR levels will be determined by the suPARnostic TurbiLatex quantitative turbidimetric immunoassay (ViroGates A/S, Denmark), also on the Architect c8000 automatic analytical system.
  Other Names: Soluble Urokinase Plasminogen Activator Receptor

SUMMARY:
The purpose of the study is to recognize the diagnostic and/or prognostic value of IMA, as It reflects the degree of ischemia regardless of the affected organ.

Our sample, which will be taken from the Pulmonology/Covid-19 Department and the Outpatient Clinic of the Pulmonology Department of University Hospital of Larissa, will be divided into two groups. The first group will be the study group, which will include patients with confirmed COVID-19 infection, while the second group will be the control group, which will include healthy volunteers. From the study population will be collected demographics, medical history, medication, symptoms, vital points, arterial blood gases, viral load from RT-PCR for SARS-COV2 and findings from imaging and laboratory assessment. On a daily basis, during their treatment, their vital points, their laboratory tests and the presence of possible complications will be recorded.

Expected results are: 1) Comparison of IMA levels between COVID-19 patients and healthy volunteers, 2) The IMA contribution, during their admission to the hospital, to the prediction of the risk of deterioration and severe respiratory failure, 3) The increase of the predictive accuracy of SuPAR as a risk stratification biomarker, after its combination with IMA, 4) The estimation of IMA on the 10th day of illness in patients with severe respiratory failure, 5) The possibility of predicting with greater accuracy the probability of admission to the ICU, by measuring the IMA on the 10th day of illness compared to the IMA of admission.

DETAILED DESCRIPTION:
Endothelial activation and dysfunction are associated with COVID-19 severity. Epidemiological studies suggest that severe cases or deaths due to COVID-19 frequently present with underlying comorbidities, such as advanced age, hypertension, diabetes, and cardiovascular diseases. Endothelial dysfunction, with the subsequent use of the complement, the hypercoagulable state and production of thrombin appears to be the common denominator of varieties of clinical signs and symptoms of COVID-19, which are directly associated with thromboembolic events. Necropsy findings in patients with COVID-19 have shown catastrophic microvascular injury, with pulmonary endotheliitis, thrombosis and angiogenesis being distinct pathophysiological features of the lungs in patients with COVID-19 compared with H1N1 patients and uninfected controls.

Venous thromboembolic disease, which can manifest as Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE), often occurs in patients with severe COVID-19, despite prophylactic anticoagulation. PE has been found in almost 20% of patients, despite having received anticoagulant treatment. In another study, necropsy was performed in 12 patients with COVID-19, of whom were receiving anticoagulants. DVT was detected in 7 (58%) patients, although none of them had a clinical suspicion. PE was the leading cause of death in 4 patients. Venous thrombosis occurs in particularly high rates (14-81%) in critically ill COVID-19 patients admitted to Intensive Care Units (ICU). In fact, PE has been recorded as the most common thrombotic complication in these patients with a frequency of up to 81%. In hospitalized patients with COVID-19, venous thrombosis occurs less frequently (3-21%), while for outpatients there are insufficient data. In addition to DVT, cases of acute ischemia of the upper or lower extremity with a potential need for surgery have also been reported as a less common arterial thrombotic complication in COVID-19.

In addition, acute myocardial ischemia is the most commonly reported cardiovascular complication of COVID-19. The prevalence of myocardial ischemia varies from 7% to 28%. Studies have correlated the increase in troponin in hospitalized patients with a more severe clinical course and worse prognosis.

Ischemic stroke is another common extrapulmonary thromboembolic complication of COVID-19. There are reports of ischemic stroke as the first symptom of infection (appearing especially as a middle cerebral artery thrombosis, even in young patients) and as a complication during hospitalization. In retrospective observational studies, the prevalence of ischemic stroke in this population ranges from 1.3% to 46%. The most likely mechanism of strokes during COVID-19 is considered to be subsequent hypercoagulability and vascular endothelial dysfunction through activation of inflammatory cytokines.

Human serum albumin is a peptide, which consists of 585 amino acids bonded in a specific sequence in humans. The ischemia modified albumin (IMA) molecule was identified in early 2000s, when it was observed that hypoxic-induced ischemia resulted in a modification in the circulating albumin molecule. Under ischemic conditions, the N-terminus of albumin is differentiated, possibly as a result of hypoxia, oxidation, free radicals and energy-dependent changes in membranes. This modification at the N-terminus of albumin can be indirectly evaluated. When cobalt (in vitro) is added to an ischemic sample, normal albumin molecules will bind to it, leaving a small percentage free, while IMA cannot bind to the added cobalt due to its modification at its binding site. Elevated IMA percentages result in more unbound cobalt, which can be detected by the addition of a chromatographic agent, such as dithiothreitol, and evaluated photospectrometrically. The increase of IMA is inversely related to the amount of cobalt, which causes an increase in the colour product. This is the basis of the Albumin Cobalt - Binding test, ACB test.

IMA has been studied as an indicator of cardiac ischemia but has also been found increased in patients with endothelial dysfunction, infections and sepsis. It also increases in patients with cerebral ischemia, pulmonary embolism, deep vein thrombosis, heart failure, intestinal ischemia etc. IMA values have a normal distribution in the control population and are not related to age and gender. IMA, which is the only ischemia biomarker that has reached the level of clinical evaluation, increases within a few minutes of the onset of ischemia regardless of the affected organ-tissue.

SuPAR (Soluble urokinase Plasminogen Activating Receptor) is the soluble form of uPAR, a protein that is primarily expressed in cells of the immune system, including neutrophils, activated T-lymphocytes, and macrophages. The uPAR binds to the cell membrane with a glycosylphosphatidyl-inositol (GPI). When uPAR is released from the cell membrane, it becomes soluble (SuPAR) and can be measured as a stable protein in various biological fluids, such as plasma, urine and cerebrospinal fluid. SuPAR levels in healthy people are quite stable in the blood and urine. Elevated levels of SuPAR reflect the activation of the immune system and have been evaluated as an indicator of inflammation and organ damage in a few diseases, including COVID-19. Studies on the concentration of SuPAR in 57 patients with COVID-19 pneumonia, showed that SuPAR concentrations were higher in patients who eventually developed severe respiratory failure and required mechanical ventilation, compared to patients who did not develop severe respiratory failure. More specifically, concentrations greater than or equal to 6 ng/ml had a sensitivity of 85.7% to predict the adverse outcome even 12 days before happening. SuPAR appears to be an important risk stratification tool in patients with COVID-19, as it can early identify patients who will develop severe respiratory failure or that need mechanical ventilation.

Since this is the first study of IMA in patients with COVID-19, the primary aim of the study is to investigate whether IMA levels at admission or at day 10 from symptoms onset (peak of symptoms) will be higher in patients with COVID-19 pneumonia compared to healthy individuals. The secondary aim is to assess whether IMA can predict severe respiratory failure and deterioration risk and whether combination with SuPAR will increase its accuracy.

Participants: 2 study groups will be included:

i) 128 patients with confirmed COVID-19 disease (study group, group 1) ii) 64 healthy volunteers without any of the exclusion criteria (control group, group 2) Patients from the study group will be divided into two subgroups, those with severe respiratory failure (PaO2/FiO2 <150mmHg) and those without severe respiratory failure (PaO2/FiO2 >150mmHg) Furthermore, they will be divided into those with or without deterioration risk defined as need for high flow nasal cannula, mechanical ventilation, ICU admission or death.

Type of study: This will be a prospective observational study that will be carried out at the Pulmonology/Covid-19 Department of the University General Hospital of Larissa.

Power analysis: For a statistical power of 90% with a probability of α-error of 0.05 and Group 1/Group 2 ratio 2:1, it was estimated that 64 people are needed in the control group (group 2) and 128 in the study group (group 1).

Interventions: Blood samples will be collected at admission for measurement of IMA and SuPAR levels and at day 10 from symptom onset (peak of symptoms) for IMA level.

Blood sample collection: Samples will be collected in blood collection tubes containing K2EDTA as anticoagulant and serum separation gel tubes for SuPAR and IMA assays respectively. The samples will be centrifuged (at 3000 x g for 10 minutes) within the first 3 hours of sampling. Then, both plasma and serum samples will be placed in Eppendorf tubes and stored at -80oC.

IMA and SuPAR measurements: IMA levels will be determined according to the principles of the ACB assay, using the commercially available "Ischemia Modified Albumin Assay Kit" method (Abbexa LTD, Cambridge, UK), on the Architect c8000 automatic analytical system (Abbott, USA). SuPAR levels will be determined by the suPARnostic TurbiLatex quantitative turbidimetric immunoassay (ViroGates A/S, Denmark), also on the Architect c8000 automatic analytical system.

Monitoring/Recording: Demographics (age, sex, nationality), date of admission, comorbidities, medication, symptoms, vital signs (heart rate, temperature, blood pressure, respiratory rate, arterial blood oxygen saturation and PaO2/FiO2 ratio), arterial blood gases (PaO2, PaCO2, pH, HCO3), lactic acid, viral load from RT-PCR for SARS-COV2 and the findings from the imaging and laboratory test (hemoglobin, hematocrit, white blood cells, neutrophils, lymphocytes, platelets, PT, INR, aPTT, fibrinogen, d-dimers, CRP, ferritin, LDH, troponin, urea, creatinine, AST, ALT, ALP, CPK, potassium, sodium, calcium, total protein, albumin, total bilirubin) will be recorded on admission.

Vital signs (heart rate, temperature, blood pressure, respiratory rate, arterial blood oxygen saturation and PaO2/FiO2 ratio), laboratory findings (as mentioned above) and the presence of any complications (pneumonia, ARDS, pulmonary embolism, stroke, acute renal failure, multiorgan failure, arrhythmias, shock, pseudomembranous colitis, etc.) will be recorded daily.

Expected results: i) IMA levels are expected to be higher in patients with COVID-19 compared to healthy volunteers ii) IMA levels at admission are expected to be higher in patients that will develop severe respiratory failure or with deterioration risk iii) IMA levels at day 10 from symptom onset are expected to be higher in patients with severe respiratory failure and predict deterioration risk with a greater accuracy iv) SuPAR levels are expected to be higher in patients with COVID-19 compared to healthy volunteers v) SuPAR levels at admission are expected to be higher in patients that will develop severe respiratory failure or with deterioration risk vi) Combination of IMA and SuPAR, is expected to increase the predictive accuracy of SuPAR

To our knowledge, this will be the first study of Ischemia Modified Albumin in patients with COVID-19. Prognosis is a key driver of clinical decision-making. If the correlation between IMA levels and poor prognosis is proved, it will become a useful tool for the risk stratification of COVID-19 patients. Furthermore, the combination of an ischemia biomarker, such as IMA, with an inflammatory biomarker, like SuPAR might be the key to this approach.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Positive nasopharyngeal test for SARS-CoV-2 confirmed by RT-PCR

Exclusion Criteria:

* Age < 18 years old
* SARS-CoV-2 infection not confirmed by RT PCR
* No consent for participation in the study
* Acute ischemic disease prior to SARS-CoV-2 (trauma, mesenteric ischemia, stroke, liver disease, venous thromboembolic disease, acute coronary syndrome in the last 3 months, etc.)
* Pregnancy
* Immunosuppression
* Albumin < 2gr/dl or > 5.5gr/dl

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who are admitted to the Hospital due to Covid-19
Sampling Method: Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Hospitalization outcome | Up to 8 weeks
  Admission to ICU, death, discharge

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios D. Pagonis, Resident, Principal Investigator — University Hospital of Larissa, Pulmonology Department
Locations (1):
- Larissa University Hospital, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Background] Steinberg BE, Goldenberg NM, Lee WL. Do viral infections mimic bacterial sepsis? The role of microvascular permeability: A review of mechanisms and methods. Antiviral Res. 2012 Jan;93(1):2-15. doi: 10.1016/j.antiviral.2011.10.019. Epub 2011 Nov 2. PMID 22068147
- [Background] Goeijenbier M, van Wissen M, van de Weg C, Jong E, Gerdes VE, Meijers JC, Brandjes DP, van Gorp EC. Review: Viral infections and mechanisms of thrombosis and bleeding. J Med Virol. 2012 Oct;84(10):1680-96. doi: 10.1002/jmv.23354. PMID 22930518
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Menter T, Haslbauer JD, Nienhold R, Savic S, Hopfer H, Deigendesch N, Frank S, Turek D, Willi N, Pargger H, Bassetti S, Leuppi JD, Cathomas G, Tolnay M, Mertz KD, Tzankov A. Postmortem examination of COVID-19 patients reveals diffuse alveolar damage with severe capillary congestion and variegated findings in lungs and other organs suggesting vascular dysfunction. Histopathology. 2020 Aug;77(2):198-209. doi: 10.1111/his.14134. Epub 2020 Jul 5. PMID 32364264
- [Background] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Cui S, Chen S, Li X, Liu S, Wang F. Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia. J Thromb Haemost. 2020 Jun;18(6):1421-1424. doi: 10.1111/jth.14830. Epub 2020 May 6. PMID 32271988
- [Background] Lodigiani C, Iapichino G, Carenzo L, Cecconi M, Ferrazzi P, Sebastian T, Kucher N, Studt JD, Sacco C, Bertuzzi A, Sandri MT, Barco S; Humanitas COVID-19 Task Force. Venous and arterial thromboembolic complications in COVID-19 patients admitted to an academic hospital in Milan, Italy. Thromb Res. 2020 Jul;191:9-14. doi: 10.1016/j.thromres.2020.04.024. Epub 2020 Apr 23. PMID 32353746
- [Background] Artifoni M, Danic G, Gautier G, Gicquel P, Boutoille D, Raffi F, Neel A, Lecomte R. Systematic assessment of venous thromboembolism in COVID-19 patients receiving thromboprophylaxis: incidence and role of D-dimer as predictive factors. J Thromb Thrombolysis. 2020 Jul;50(1):211-216. doi: 10.1007/s11239-020-02146-z. PMID 32451823
- [Background] Middeldorp S, Coppens M, van Haaps TF, Foppen M, Vlaar AP, Muller MCA, Bouman CCS, Beenen LFM, Kootte RS, Heijmans J, Smits LP, Bonta PI, van Es N. Incidence of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1995-2002. doi: 10.1111/jth.14888. Epub 2020 Jul 27. PMID 32369666
- [Background] Vacirca A, Faggioli G, Pini R, Teutonico P, Pilato A, Gargiulo M. Unheralded Lower limb threatening ischemia in a COVID-19 patient. Int J Infect Dis. 2020 Jul;96:590-592. doi: 10.1016/j.ijid.2020.05.060. Epub 2020 May 22. PMID 32447121
- [Background] Kaur P, Qaqa F, Ramahi A, Shamoon Y, Singhal M, Shamoon F, Maroules M, Singh B. Acute upper limb ischemia in a patient with COVID-19. Hematol Oncol Stem Cell Ther. 2021 Dec;14(4):348-350. doi: 10.1016/j.hemonc.2020.05.001. Epub 2020 May 13. PMID 32405288
- [Background] Bansal M. Cardiovascular disease and COVID-19. Diabetes Metab Syndr. 2020 May-Jun;14(3):247-250. doi: 10.1016/j.dsx.2020.03.013. Epub 2020 Mar 25. PMID 32247212
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Clerkin KJ, Fried JA, Raikhelkar J, Sayer G, Griffin JM, Masoumi A, Jain SS, Burkhoff D, Kumaraiah D, Rabbani L, Schwartz A, Uriel N. COVID-19 and Cardiovascular Disease. Circulation. 2020 May 19;141(20):1648-1655. doi: 10.1161/CIRCULATIONAHA.120.046941. Epub 2020 Mar 21. PMID 32200663
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 31;368:m1295. doi: 10.1136/bmj.m1295. No abstract available. PMID 32234718
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Avula A, Nalleballe K, Narula N, Sapozhnikov S, Dandu V, Toom S, Glaser A, Elsayegh D. COVID-19 presenting as stroke. Brain Behav Immun. 2020 Jul;87:115-119. doi: 10.1016/j.bbi.2020.04.077. Epub 2020 Apr 28. PMID 32360439
- [Background] Oxley TJ, Mocco J, Majidi S, Kellner CP, Shoirah H, Singh IP, De Leacy RA, Shigematsu T, Ladner TR, Yaeger KA, Skliut M, Weinberger J, Dangayach NS, Bederson JB, Tuhrim S, Fifi JT. Large-Vessel Stroke as a Presenting Feature of Covid-19 in the Young. N Engl J Med. 2020 May 14;382(20):e60. doi: 10.1056/NEJMc2009787. Epub 2020 Apr 28. No abstract available. PMID 32343504
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Varatharaj A, Thomas N, Ellul MA, Davies NWS, Pollak TA, Tenorio EL, Sultan M, Easton A, Breen G, Zandi M, Coles JP, Manji H, Al-Shahi Salman R, Menon DK, Nicholson TR, Benjamin LA, Carson A, Smith C, Turner MR, Solomon T, Kneen R, Pett SL, Galea I, Thomas RH, Michael BD; CoroNerve Study Group. Neurological and neuropsychiatric complications of COVID-19 in 153 patients: a UK-wide surveillance study. Lancet Psychiatry. 2020 Oct;7(10):875-882. doi: 10.1016/S2215-0366(20)30287-X. Epub 2020 Jun 25. PMID 32593341
- [Background] Romero-Sanchez CM, Diaz-Maroto I, Fernandez-Diaz E, Sanchez-Larsen A, Layos-Romero A, Garcia-Garcia J, Gonzalez E, Redondo-Penas I, Perona-Moratalla AB, Del Valle-Perez JA, Gracia-Gil J, Rojas-Bartolome L, Feria-Vilar I, Monteagudo M, Palao M, Palazon-Garcia E, Alcahut-Rodriguez C, Sopelana-Garay D, Moreno Y, Ahmad J, Segura T. Neurologic manifestations in hospitalized patients with COVID-19: The ALBACOVID registry. Neurology. 2020 Aug 25;95(8):e1060-e1070. doi: 10.1212/WNL.0000000000009937. Epub 2020 Jun 1. PMID 32482845
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Bar-Or D, Lau E, Winkler JV. A novel assay for cobalt-albumin binding and its potential as a marker for myocardial ischemia-a preliminary report. J Emerg Med. 2000 Nov;19(4):311-5. doi: 10.1016/s0736-4679(00)00255-9. PMID 11074321
- [Background] Pantazopoulos I, Papadimitriou L, Dontas I, Demestiha T, Iakovidou N, Xanthos T. Ischaemia modified albumin in the diagnosis of acute coronary syndromes. Resuscitation. 2009 Mar;80(3):306-10. doi: 10.1016/j.resuscitation.2008.10.035. Epub 2008 Dec 25. PMID 19111377
- [Background] Kaya Z, Kayrak M, Gul EE, Altunbas G, Toker A, Kiyici A, Gunduz M, Alibasic H, Akilli H, Aribas A. The role of ischemia modified albumin in acute pulmonary embolism. Heart Views. 2014 Oct-Dec;15(4):106-10. doi: 10.4103/1995-705X.151083. PMID 25774252
- [Background] Park J, Ahn S, Lee S, Song J, Moon S, Kim J, Cho H. Association of ischemia modified albumin with mortality in qSOFA positive sepsis patients by sepsis-3 in the emergency department. Am J Emerg Med. 2021 Jun;44:72-77. doi: 10.1016/j.ajem.2021.01.059. Epub 2021 Jan 29. PMID 33582611
- [Background] Choo SH, Lim YS, Cho JS, Jang JH, Choi JY, Choi WS, Yang HJ. Usefulness of ischemia-modified albumin in the diagnosis of sepsis/septic shock in the emergency department. Clin Exp Emerg Med. 2020 Sep;7(3):161-169. doi: 10.15441/ceem.19.075. Epub 2020 Sep 30. PMID 33028058
- [Background] Menon B, Ramalingam K, Krishna V. Study of Ischemia Modified Albumin as a Biomarker in Acute Ischaemic Stroke. Ann Neurosci. 2018 Dec;25(4):187-190. doi: 10.1159/000488188. Epub 2018 Jun 28. PMID 31000956
- [Background] Balamir I, Ates I, Topcuoglu C, Turhan T. Association of Endocan, Ischemia-Modified Albumin, and hsCRP Levels With Endothelial Dysfunction in Type 2 Diabetes Mellitus. Angiology. 2018 Aug;69(7):609-616. doi: 10.1177/0003319717740781. Epub 2017 Nov 26. PMID 29172652
- [Background] Balta S. Endothelial Dysfunction and Inflammatory Markers of Vascular Disease. Curr Vasc Pharmacol. 2021;19(3):243-249. doi: 10.2174/1570161118666200421142542. PMID 32316894
- [Background] Chalkias A, Mouzarou A, Samara E, Xanthos T, Ischaki E, Pantazopoulos I. Soluble Urokinase Plasminogen Activator Receptor: A Biomarker for Predicting Complications and Critical Care Admission of COVID-19 Patients. Mol Diagn Ther. 2020 Oct;24(5):517-521. doi: 10.1007/s40291-020-00481-8. PMID 32613288
- [Background] Rovina N, Akinosoglou K, Eugen-Olsen J, Hayek S, Reiser J, Giamarellos-Bourboulis EJ. Soluble urokinase plasminogen activator receptor (suPAR) as an early predictor of severe respiratory failure in patients with COVID-19 pneumonia. Crit Care. 2020 Apr 30;24(1):187. doi: 10.1186/s13054-020-02897-4. No abstract available. PMID 32354367